CLINICAL TRIAL: NCT06781125
Title: A Phase I Clinical Trial to Evaluate the Safety and Tolerability of JCXH-211 Intratumoral Injection Combined With Anti-PD-1 Antibody IV Infusion in Patients With Malignant Solid Tumors
Brief Title: One Trial of JCXH-211 Intratumoral Injection Combined With Anti-PD-1 Antibody in Patients With Malignant Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Immorna Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JCXH-211-006
Record Dates: First submitted 2024-11-12; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Malignant Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phase Ia will be planned in 2 dose groups, Phase Ib will select the optimal dose based Phase Ia (Experimental)
  Interventions: Drug: JCXH-211 Intratumoral Injection Combined with Anti-PD-1 Antibody IV infusion

INTERVENTIONS:
Drug: JCXH-211 Intratumoral Injection Combined with Anti-PD-1 Antibody IV infusion — JCXH-211:Tumor lesions are selected for intratumoral injection, and target or non-target lesions can be selected. The number of lesions selected for injection will be at the investigator 's discretion based on the patient' s general condition and tolerability .
  Anti-PD-1 antibody:Dosage and administration according to the instructions.

SUMMARY:
This is an open-label, dose-escalation and dose-expansion Phase I clinical study divided into Phase Ia and Phase Ib to evaluate the safety and tolerability of JCXH-211 combined with anti-PD-1 antibody in patients with malignant solid tumors.

DETAILED DESCRIPTION:
Phase Ia: Dose escalation study of intratumoral injection of JCXH-211 combined with anti-PD-1 antibody IV infusion A dose escalation study of intratumoral injection of JCXH-211 combined with anti-PD-1 antibody IV infusion will be planned in 2 dose groups . Three to six patients will be enrolled in each dose group.

Phase Ib:Dose Expansion Study of JCXH-211 Combined with Anti-PD-1 Antibody In this part of the study, the sponsor and investigator select the optimal dose based on the safety, PK, PD and preliminary efficacy results of the dose escalation phase, and select 1 to 2 of the tumors for JCXH-211 combined with anti-PD-1 antibody dose expansion study with reference to the approved indications of anti-PD-1 antibody (Toripalimab ) in China, and planned to enroll 15 to 30 patients in each cohort of combination therapy.

Tumor response assessments will be performed using RECIST1.1 and iRECIST at the end of study treatment/early withdrawal visit and every 6 weeks during treatment.

All patients will be followed for safety and survival. The data cut-off date for study is defined as 6 months after the last patient is enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, aged 18 to 75 years;
2. patients with malignant solid tumors confirmed by pathology and/or cytology who have progressed or are intolerant to standard treatment (except best supportive care); Including patients who have received prior anti-PD-1 antibody therapy; patients who have been approved as eligible for Toripalimab:
3. General condition score ECOG 0 ~ 1;
4. Expected survival of more than 3 months;

Exclusion Criteria:

1. Known or suspected allergy to the ingredients of the study drug or its analogues; allergic history to another monoclonal antibody;
2. patients who have previously received IL-12 therapy (alone or as part of a treatment regimen), except those who have participated in tolerance to a single intratumoral injection;
3. patients who have previously received treatment with anti-PD-1, anti-PD-L1, or anti-PD-L2 agents, or have received treatment directed at another stimulatory or coinhibitory T-cell receptor (e.g., CTLA-4, OX-40, CD137), and discontinued treatment due to Grade 3 or higher immune-related adverse events (irAEs);

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-02-10 (Estimated); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | The DLT observation period is 28 days after first dose of JCXH-211 combined with anti-PD-1 antibody

CONTACTS AND LOCATIONS:
Overall Officials: RuiHua Xu, Principal Investigator — Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No